CLINICAL TRIAL: NCT06453486
Title: Ablative Radiation Therapy With High Dose Geometric Boost for Locally Advanced Pancreatic Cancer Patients Following Treatment Response Evaluation of Standard of Care Induction Chemotherapy (ABLATE): a Phase II Clinical Trial
Brief Title: A Study of High Dose Radiation Therapy for Locally Advanced Pancreatic Cancer That Responded to Initial Chemotherapy Treatment
Acronym: ABLATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-031
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: High dose radiation therapy — High dose radiation refers to the administration of a concentrated beam of radiation to target and treat the tumor. High dose radiation therapy typically involves delivering radiation in fractions over a set period. For instance, options such as:
  * 50Gy/5Fx: 50 Gray delivered over 5 fractions, administered every other day over 2 weeks.
  * 67.5Gy/15Fx: 67.5 Gray delivered over 15 fractions, administered once a day over 3 weeks.
  * 75Gy/25Fx: 75 Gray delivered over 25 fractions, administered once a day over 5 weeks.
  These numbers denote the total dose of radiation (in Gray, abbreviated as Gy) delivered over a specific number of fractions (abbreviated as Fx), and the respective time frames for administration. The selection of radiation therapy (RT) dose levels for participants is guided by the expertise and evaluation of the radiation oncologist.

SUMMARY:
The goal of this clinical trial is to test the effect of high-dose radiation therapy after initial chemotherapy in patients with locally advanced pancreatic cancer. The main question it aims to answer is:

• For patients with locally advanced pancreatic cancer that responded to initial chemotherapy (stayed stable or decreased in size), will high-dose RT (radiation therapy) contribute to improving treatment outcomes, enhancing quality of life, or increasing overall survival rates?

Participants will:

* Undergo an optional tumor biopsy.
* Be treated with high dose radiation therapy.
* Complete quality of life questionnaires.
* Donate research blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological or cytological diagnosis of LAPC.
* Have pancreatic tumour <8.0 cm in greatest axial dimension at the time of treatment planning but final determination of eligibility will be based upon satisfying the radiation normal tissue constraints.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Karnofsky ≥70%).
* Life expectancy of greater than 6 months, as judged by the investigator.
* Patients must have had prior first-line chemotherapy for this cancer for at least 16 weeks without clinical or radiographic progression. There should be a washout of at least 2 weeks from first-line chemotherapy and start of therapy on clinical trial.
* Ability to understand and willing to sign a written informed consent document.
* Women must not be pregnant or breast-feeding. All females of child bearing potential must have a serum or urine pregnancy test to rule out pregnancy within 4 weeks prior to registration. All breastfeeding women should discontinue breastfeeding prior to study registration.

Exclusion Criteria:

* Metastatic disease at the time of registration
* Age<18.
* Patients who have had prior systemic treatment (chemotherapy or any other anti-cancer agent) in the metastatic setting.
* Prior radiotherapy to the upper abdomen region that would result in overlap of RT volume for the current study.
* Patients who are currently on anti-cancer treatment including chemotherapy.
* Uncontrolled inter-current illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and breastfeeding women.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Individuals with a history of a different malignancy except if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Individuals with diseases precluding high dose ablative RT (e.g. scleroderma, gastric or bowel ulceration or perforation within the planned irradiated volume)
* Patient should NOT be treated with MR-Linac if they have any contraindications for MRI, including presence of a heart pacemaker, (ferrous) metallic foreign bodies, and severe claustrophobia. Patients will be screened and excluded from the study if they have previous anaphylactic reactions to gadolinium and severe kidney disease (glomerular filtration rate < 30mL/min/1.73m2) or acute kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  To evaluate the efficacy of ablative radiation therapy with high dose geometric boost for patients with locally advanced pancreatic cancer with stable disease or partial response following standard of care induction chemotherapy, as measured by median overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Erica Tsang, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No